CLINICAL TRIAL: NCT03754010
Title: Evaluation of Clinical and Biochemical Effects of Hyaluronic Acid on Periodontitis: A Split-mouth Randomized-controlled Trial
Brief Title: Does Hyaluronic Acid Affect Periodontal Treatment?
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Hacer Sahin Aydinyurt, Assist Prof, Yuzuncu Yil University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 19.07.2017/09
Record Dates: First submitted 2018-11-15; First posted 2018-11-27 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Periodontitis
Keywords: periodontitis; hyaluronic acid; scaling and root planning; adenosione deaminase; catalase; glutathione
MeSH Terms: conditions — Periodontitis | interventions — Tooth Exfoliation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Scaling and root planning (SRP) (Placebo Comparator): Under local anesthesia, full-mouth SRP was performed within 24 h in a single or two sessions using ultrasonic and hand instruments (Gracey, Hu-Friedy, Chicago, IL, USA) by a single investigator (DA). Immediately after the SRP, HA gel (Gengigel, Hyaluronic acid, gingival gel, Ricefarma S.R.L, Italy) or mouthrinse was performed according to the groups' procedure. In Group 1, the periodontal sulcus was irrigated with saline solution after SRP.
  Interventions: Procedure: Scaling and root planning
- Hyaluronic acid gel (HA) and SRP (Experimental): Group 2, after SRP was performed and irrigated with saline the area was dried with a soft air and, then, a gel containing HA was applied intrasulcular.
  Interventions: Procedure: Scaling and root planning; Drug: Hyaluronic acid gel (HA) and SRP
- HA mouthrinse and SRP (Experimental): In Group 3, HA hydrogel mouthrinse (Gengigel, Hyaluronic acid, Hydrogel moutrinse for gums, Ricefarma S.R.L, Italy) were used as an irrigator after SRP.
  Interventions: Procedure: Scaling and root planning; Drug: HA mouthrinse and SRP
- HA mouthrinse+gel and SRP (Experimental): In Group 4, after SRP was performed, the sulcus was irrigated with HA hydrogel mouthrinse and, then, intrasulculary HA gingival gel was applied.
  Interventions: Procedure: Scaling and root planning; Drug: HA mouthrinse+gel and SRP

INTERVENTIONS:
Procedure: Scaling and root planning — Under local anesthesia, full-mouth SRP will be performed by a single investigator. Immediately after the SRP, HA gel or mouthrinse will perform according to the groups' procedure. In Group 1, the periodontal sulcus will be irrigated with saline solution after SRP.
Drug: Hyaluronic acid gel (HA) and SRP — In Group 2, after SRP will be performed and irrigated with saline the area was dried with a soft air and, then, a gel containing HA will be applied intrasulcular.
  Other Names: HA and SRP
  Arms: Hyaluronic acid gel (HA) and SRP
Drug: HA mouthrinse and SRP — In Group 3, HA hydrogel mouthrinse will be used as an irrigator after SRP.
  Other Names: HAmo+SRP
  Arms: HA mouthrinse and SRP
Drug: HA mouthrinse+gel and SRP — In Group 4, after SRP will be performed, the sulcus was irrigated with HA hydrogel mouthrinse and, then, intrasulculary HA gingival gel will be applied.
  Other Names: HAmo+HAgel+SRP
  Arms: HA mouthrinse+gel and SRP

SUMMARY:
Objective: The aim of this study is to evaluate the effect of HA as an adjunct to scaling and root planning (SRP) on clinical parameters, periodontal inflamed surface area (PISA) and adenosine deaminase (ADA), catalase (CAT), and glutathione (GSH) levels in gingival crevicular fluid (GCF) in patients with periodontitis.

DETAILED DESCRIPTION:
Design: A total of 24 Stage II-III periodontitis patients will be included in this split-mouth, randomized-controlled study. The study population will be divided into four groups: in Group 1 (SRP): SRP+ saline; in Group 2 (SRP+HAgel): SRP + HA gel; in Group 3 (SRP+HAmo): SRP+ HA mouthrinse; and in Group 4 (SRP+HAmo+HAgel): SRP+HA mouthrinse + HA gingival gel were applied. At baseline and Week 4 periodontal clinical parameters and PISA will be calculated. Also, GCF amount will be collected to evaluate ADA, CAT, and GSH by spectrophotometric analysis.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy
* moderate-to-severe periodontitis
* at least five sites with ≥5mm probing depth (PD)
* at least ≥20 teeth
* Stage II-III periodontitis according to the 2017 World Workshop
* Age between18-55

Exclusion Criteria:

* receiving systemic or local antibiotics within the past six months
* prior surgical or non-surgical periodontal treatment within the past six months
* smoking
* pregnancy
* lactation
* age ≤18 years or ≥55 years
* hypertension
* known chronic systemic diseases (i.e., diabetes mellitus, rheumatoid arthritis), - - known hypersensitivity to one of the ingredients of the HA preparation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
plaque index | Change from Baseline to week 4
  in accordance with the Sillness and Löe index (Silness & Löe, 1964)
gingival index (GI) | Change from Baseline to week 4
  confirming to Silness and Löe index (Löe & Silness, 1963)
bleeding on probing (BOP) | Change from Baseline to week 4
  according to Ainoma and Bay (AINAMO & Bay, 1975);
Probing depth (PD) | Change from Baseline to week 4
  as the measurement of the length between the bottom of the periodontal pocket to marginal gingiva;
gingival recession height (GRH) | Change from Baseline to week 4
  as the measurement of the distance between the marginal gingiva and cemento-enamel junction
clinical attachment level (CAL) | Change from Baseline to week 4
  as the sum of gingival recession height and probing depth will be recorded.

SECONDARY OUTCOMES:
Changes of Periodontal inflammed surface area | Change from Baseline Baseline to week 4
  All clinical parameters will be entered on Microsoft Excel Program (www.parsprototo.info) which constructed for calculating PISA. The BOP percentage for each tooth will be calculated by entering "number sites with BOP" values in the Excel program.
Changes of Adenosine deaminase (ADA) levels in gingival crevicular fluid | Changes from Baseline to week 1,2,4
  The ADA activity will be evaluated spectrophotometrically
Changes of Catalase levels in gingival crevicular fluid | Changes from Baseline to week 1,2,4
  The catalase activity will be evaluated spectrophotometrically
Changes of Glutathione levels in gingival crevicular fluid | Changes from Baseline to week 1,2,4
  The Glutathione activity will be evaluated spectrophotometrically

CONTACTS AND LOCATIONS:
Overall Officials: Hacer Sahin Aydinyurt, Assist Prof, Study Director — Yuzuncu Yil University
Locations (1):
- Van Yuzuncu Yil University Faculty of Dentistry, Van, Turkey (Türkiye)

REFERENCES:
- [Derived] Aydinyurt HS, Akbal D, Altindal D, Bozoglan A, Ertugrul AS, Demir H. Evaluation of biochemical and clinical effects of hyaluronic acid on non-surgical periodontal treatment: a randomized controlled trial. Ir J Med Sci. 2020 Nov;189(4):1485-1494. doi: 10.1007/s11845-020-02230-6. Epub 2020 May 21. PMID 32436173